CLINICAL TRIAL: NCT01432288
Title: Effects of Touch and Attention on Central Nervous System Resting State Network (RSN) Activity
Brief Title: Touch and Attention MRI Study
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: WFUIRB00016834
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will measure resting state network central nervous system activity by functional magnetic resonance imaging (fMRI) during 4 separate interactions with a clinician. 1.

Hypothesis 1. Because they are different sensory systems, there will be different patterns of Mirror Neuron System (MNS)and Resting State Network (RSN) Central Nervous System (CNS) activity for visual vs. tactile stimulation, regardless of Loving Kindness Meditation (LKM).

Hypothesis 2. Because of unconscious, non-verbal signals, such as the practitioner's facial expression and respiratory rate, subjects' patterns of MNS and RSN CNS activity will differ for LKM+ vs. LKM- stimulation for both visual and tactile interventions.

Hypothesis 3. Because there is greater opportunity to detect signals from two sensory systems than one, the differences between CNS MNS and RSN activity patterns for LKM+ and LKM- will be greater for combined visual + tactile than for either visual or tactile stimulation alone.

DETAILED DESCRIPTION:
This project builds on our previous research to build a platform for a successful NIH proposal to address a key gap in our understanding of the mechanism of non-verbal clinician-patient communication on physiology and behavior. Social neuroscience is a rapidly growing area of research that offers unique opportunities to better understand the mechanisms underlying common observations about clinician-patient interactions.The purpose of this study is to better understand the CNS mechanisms underlying the observed changes in self-reported well-being and ANS activity by evaluating resting fMRI activity under controlled conditions. The specific aims are to compare resting fMRI activity in the mirror neuron system (MNS) and resting state networks (RSN), reflected specifically in the Insula, Anterior Cingulate Cortex (ACC), Precuneus, Posterior Cingulate Cortex (PCC), Amygdala, Bilateral Inferior Parietal Cortex, Primary Motor-Visual System, and Dorsal Medulla while viewing touch with lovingkindness meditation lovingkindness meditation vs no lovingkindness meditation, receiving touch with lovingkindness meditation vs no lovingkindness meditation and both viewing and receiving touch with lovingkindness meditation vs no lovingkindness meditation. This is a descriptive study to generate sample size estimates for an NIH RO1 proposal.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* healthy
* can understand and respond to verbal directions while in an MRI

Exclusion Criteria:

* blind
* undergone treatment for brain tumor, stroke, intracranial hemorrhage
* diabetes or any other form of peripheral neuropathy
* require a pacemaker, insulin pump or other electronic equipment
* taking beta blocking medications, systemic steroid medications or other medications likely to affect autonomic or central nervous system function

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be healthy individuals, 18< 40 years old, and can understand and respond to verbal directions while in an fMRI. Individuals over the age of 40 are excluded to provide a more homogeneous sample, to make this sample comparable to other research conducted at this institution and to decrease abnormalities in the outcome measures due to age-related changes.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathi Kemper, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Center for Biomolecular Imaging and Center for Integrative Medicine, Wake Forest University, Winston-Salem, North Carolina, United States